CLINICAL TRIAL: NCT00101699
Title: Influence of Soy Consumption on Menopause
Brief Title: Effects of Soy Consumption on Symptoms of Menopause
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: F31AT001041-01 (NIH)
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2005-01

CONDITIONS: Menopause
Keywords: Women; Soy Foods; Middle Aged

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to examine the way soy consumption affects menopausal symptoms in middle-aged Japanese women.

DETAILED DESCRIPTION:
For the past 20 years, Japanese women have reported fewer menopausal symptoms than their North American counterparts. One explanation for the disparity is the differences in diet. Evidence suggests that Japanese women consume large amounts of soy, a phytoestrogen that is structurally similar to the hormone estrogen. However, there is a lack of menopause-related research data from non-Western populations. This study will be a long-term observation of the effects of soy consumption in menopausal Japanese women.

This study will last 6 months. Participants will complete a dietary log and a menopausal symptom checklist daily. There will be three or four study visits. During these visits, participants will complete a diet questionnaire, have a blood sample collected, and be interviewed about their menopausal symptoms. Six months after study completion, participants will be sent a questionnaire about any recent menopausal symptoms they may have experienced.

ELIGIBILITY:
Inclusion Criteria:

* Japanese resident
* Menopausal

Exclusion Criteria:

* Hysterectomy, removal of ovaries, or tubal ligation with subsequent menstrual changes
* Hormones for menopause or birth control pills within 5 years of study entry
* Recent major illness
* Medication that could affect naturally-produced hormones

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2001-11; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Melissa K. Melby, MPhil, MA, Principal Investigator — Emory University
Locations (2):
- Japan (2):
  - Loma Linda Clinic, Kōriyama, Fukushima
  - Kyoto Prefectural University of Medicine, Kamigyō-ku, Kyoto